CLINICAL TRIAL: NCT04163367
Title: Can Children be Protected Against Violence and Violations From Parents? A Randomized Controlled Study of Safer Kids: A Manualized Intervention to Prevent Child Abuse
Brief Title: A Randomized Controlled Study of Safer Kids: A Manualized Intervention to Prevent Child Abuse
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Martin Forster, Principal Investigator, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Tryggare barn RCT
Record Dates: First submitted 2019-10-25; First posted 2019-11-14 (Actual); Last update posted 2025-05-20 (Actual); Status verified 2025-05

CONDITIONS: Child Abuse; Child Maltreatment
Keywords: Parenting; Randomized controlled trial; Parent-Child relations; Social services; Prevention
MeSH Terms: interventions — Methods

STUDY DESIGN:
Intervention Model Description: Participants are randomized to the control condition (intervention as usual) or the experimental condition (intervention as usual + Safer Kids - manualized parent training)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention as usual (Active Comparator): The social services standard process for families reported for violence or abuse towards children. The standard process always includes a formal investigation of the suspected violence/abuse. The investigation may or may not result in voluntary or mandatory interventions, such as family support or parent training.
  Interventions: Other: Intervention as usual (IAU)
- Intervention as usual + Safer Kids (Experimental): The procedure in this arm is exactly the same as in the active comparator arm (i.e., investigation that may be followed by interventions). In addition, the general parent training program Safer Kids is offered during the investigation to all participants in this arm.
  Interventions: Behavioral: Safer Kids; Other: Intervention as usual (IAU)

INTERVENTIONS:
Behavioral: Safer Kids — A behaviorally based parent training program with the purpose to reduce or prevent child abuse.
  Arms: Intervention as usual + Safer Kids
Other: Intervention as usual (IAU) — Everything that's included in the social service units' regular handling of cases; such as the formal investigation and family treatment. The units cannot offer Safer Kids as a part of IAU.

SUMMARY:
One of the most important responsibilities for the social services is to investigate suspected child abuse and to offer suitable intervention for the families. The lack of published studies on the effect of such interventions is therefore noteworthy. Globally, few controlled studies have been published and none of them have been conducted in Sweden. To better guide the social services in the selection of interventions, the need for Swedish studies with experimental design is therefore apparent. Previous experience in using manualized interventions with families within the social services points to the importance of regarding issues of implementation and dissemination. Interventions need to be developed and adjusted to optimize the chance of engaging families that often live under strong social pressure. The interventions also need to be designed to enable implementation and sustainability in regular services.

Safer Kids is a manualized intervention offered to caregivers under investigation for child abuse. The intervention was developed by the City of Stockholm in cooperation with practitioners within the social services. The content is based on the established parenting program Comet, but has been adjusted to suit the target group. Safer Kids has already been offered for a couple of years within the social services, but has not yet been evaluated.

In this project, a study of intervention effects will be conducted. Caregivers will be randomized to either receive Intervention as usual (IAU), or IAU plus Safer Kids. Effects on established risk-factors for child abuse, as well as the abused childrens' experiences, will be measures. Information on additional reports to the social services on child abuse will be collected, up to 30 month after the intervention.

DETAILED DESCRIPTION:
BACKGROUND:

International studies have shown prevalence rates of child abuse globally, with around 20 percent of all children being exposed to violent or abusive parenting (Stoltenborgh, Bakermans Kranenburg, Ijzendoorn, & Alink, 2013). A Swedish study showed that 15 percent of children living in Sweden sometime had experienced physical violence from a parent or close relative, from which half had been exposed several times (Annerbäck, Wingren, Svedin, & Gustafsson, 2010). Apart from the suffering caused by the abuse in itself, does the experience of child abuse act as a risk-factor for future problems. It has for example been shown that children who have experienced child abuse run a greater risk for developing depression, anxiety disorders, eating disorders, conduct disorders and substance abuse problems (Norman et al., 2012).

Despite the apparent need for effective interventions to prevent child abuse, few well-designed studies of intervention effects have been published. In a recent meta-analysis including all randomized trials of all types of interventions to prevent or treat child abuse, only 23 studies were included (Euser, Alink, Stoltenborgh, Bakermans-Kranenburg, & van IJzendoorn, 2015). The results of that analysis was also a disappointment, since the overall effect in terms of reducing or preventing child abuse was d=0.13, an effect that turned out to be non- significant after taking publication bias into account. However, a moderation analysis showed that interventions based on parent training (N=10) showed significantly larger effects than other types of interventions. In support of that result, another meta-analysis including studies of parent training interventions only, did show a significant overall effect of 11 percent absolute reduction in risk of reabuse (Vlahovicova, Melendez-Torres, Leijten, Knerr, & Gardner, 2017). Thus, even if parent training interventions show some promise, the small to non-existent intervention effects found in the meta-analyses also point to the need of developing more effective interventions.

The application of manualized interventions is rare within the social services in Sweden, but there have been a few projects in recent years with the purpose of implementing interventions that previously have been evaluated in foreign studies. One example is the iRisk-project (Broberg et al., 2015). The main purpose of that project was to investigate the ability of regular service providers to implement the interventions fith fidelity and sustainability. The effects of the interventions were also measured, but only with pre-post design without a matched control group. Both parents and the practitioners appreciated the interventions. There were also positive effects on outcome measures between pre and post the interventions, but since no matched control group was included, no safe conclusion of intervention effects could be drawn. However, several challenges were also identified in terms of implementation and sustainability. First, it was found that it was harder than expected to recruit and engage caregivers in the interventions. Secondly, several of the included service units had difficulties getting started with interventions and many reported that contacts were terminated prematurely. A third conclusion was that several practitioners described difficulties in sustaining the work with the more time consuming interventions at their service unit. A final conclusion was that practitioners found it difficult to maintain continuity in the longer interventions, due to logistic challenges for the practitioner and the families.

In summary, most previously evaluated interventions demand considerable time and resources, and there have consequently been reports of challenges in terms of implementation. In view of the prevalence of child abuse, it is therefore apparent that many families that are investigated within the services never will get access to such interventions. Furthermore, a condition in several of the existing interventions is that the suspected caregiver acknowledges the abusive act that has been committed, either in the investigation that precedes the intervention, or as a part of the intervention itself. This may pose challenges in terms of stigma and motivation to engage in the intervention. In light of these challenges, it is important to develop interventions that a) readily can be implemented with fidelity and sustainability in regular social service units, b) is less demanding and time consuming - both to be able to serve a larger number of investigated families, but also to prevent fatigue and premature termination in participating families, c) that minimize stigma and therefore can engage reluctant caregivers.

It was with some of the above challenges in mind that the City of Stockholm developed the intervention Safer Kids (Tryggare barn in Swedish), which will be evaluated in the present study. The intervention is based on the Comet program (Komet in Swedish), which is an established parenting program based on social learning theory. Practitioners at several social service units participated in the development and necessary adjustments for the target group. The program was developed in 2013-2014 and has since been implemented within the Social services and is well perceived by practitioners and caregivers, but there is no published study of its effectiveness.

PURPOSE AND RESEARCH QUESTIONS:

The purpose of this project is to evaluate the effects of Safer Kids, that is offered within the social services to caregivers suspected for child abuse. Families who are reported to the social services will be recruited and randomized to either receiving intervention as usual (IAU) or IAU plus Safer Kids. The study will answer questions pertaining possible additional effects of supplementing regular interventions with Safer kids.

The specific research questions will be:

1. What is the additional effect of Safer kids on the occurence of/time to reabuse?
2. What is the additional effect of Safer kids on established risk-factors for child abuse/reabuse?
3. What is the additional effect of Safer kids on the well-being of the abused child?
4. What is the additional effect of Safer kids on the quality of the relationship between the caregivers and the child?
5. What is the additional effect of Safer kids on the frequency of caregivers who prematurely terminates contact with the social services?
6. What is the additional effect of Safer kids on quality of life and economic outcomes?
7. How is practitioner and caregiver adherence to the Safer Kids manual related to outcomes?
8. How are practitioners and parents experiencing the feasibility of Safer Kids?

METHOD:

Participants:

Families will be recruited through the social service units that take part in the research project. Service units from all parts of Sweden are invited to the project. The following inclusion criteria were applied at the start of the project: 1) at least one caregiver in the family is suspected to have perpetrated an abusive act towards a child, 2) at least one child in the family is between 3 and 12 years old and 3) there is a decision of a formal investigation of the matter. The exclusion criterium is that families already involved in an ongoing intervention within the social services at the time of the report of the suspected act will be excluded. The inclusion and exclusion criteria were revised early during the study. For revised criteria, see the section "Eligibility".

Design:

The study is a randomized controlled trial. Families who are recruited to the study from the units who take part of the project will be randomized to either the intervention as usual at the unit (IAU) or to IAU plus Safer Kids. In the later condition, practitioners trained in Safer Kids will offer that intervention. The service units reports to the research team when a caregiver has been recruited and an assistant conducts the randomization.

The participating caregivers will answer questionnaires before the intervention, after 4 months and after 7 months. If the child participates in meetings, the practitioners will also conduct a brief interview with the child at the same time-points. Caregivers will also be asked to answer a shorter follow-up survey after 18 and 30 months. After 4, 7, 18 and 30 months from the first assessment, the practitioners will also complete a report for the research team, based on records the unit keeps for every family they have served.

Intervention:

Safer Kids was developed in 2013-2014 by the City of Stockholm. It was a joint effort between practitioners at a selected number of social service units, and researchers and developers within the City of Stockholm. The content of the program was based on the Comet program, which is a regular parent training program based on social learning theory. The Comet program has shown medium to large effects on child conduct problems in previous randomized trials (Kling, Forster, Sundell, & Melin, 2010; Stattin, Enebrink, Özdemir, & Giannotta, 2015). The intervention is delivered individually to caregivers and offered immediately after the report of suspected child abuse have reached the social services. Thus, the question of guilt for the suspected acts is not addressed with the caregiver. Instead the program is presented as a preventive effort offered to all caregivers reported to the social services, regardless of whether an investigation is started and regardless of results. The advantage with this procedure is that the practitioner can start the work with the caregivers at a moment when motivation is higher, rather than at a later point after an investigation that may take time and result in fatigue. The first step of Safer Kids is 1-3 sessions with motivational interviewing. If the caregiver decides to continue after that phase, six individual sessions with general parenting content follows (e.g., child directed play, communication skills, praise, and anger management). The six parenting sessions are followed by 1-3 follow-up sessions depending upon the need in the family. Besides the meeting with the caregiver, Safer Kids also include two individual sessions with the child (without parents if possible).

Sample size calculation:

The effects of interventions on child abuse have generally been non-existent or small (Euser et al., 2015; Vlahovicova et al., 2017). However, the effects on indirect variables (i.e., risk factors) have been in the medium range (Chen & Chan, 2016; Lundahl, Nimer, & Parsons, 2006). If an intervention should have a practical meaning, the effect sizes at least have to be between small and medium according to Cohen's standards. It was therefore decided that the sample size should be large enough to at least be able to detect effect sizes in that range. A recruitment of at least 54 families result in a statistical power of 80% to detect effect sizes of d > .35 (Faul, Erdfelder, Buchner, & Lang, 2009). This is however under optimal circumstances with no drop-out and expected heterogenity in the outcome measures. The goal is therefore set to 100 recruited families. It is expected that a rather large portion of included families will drop put, considering the high pressure and burden this group of families often experience, as well as the sensitive situation of being the subject of interventions within the social services.

Statistical analyses:

To examine possible differences between participants before the interventions, chi-squared tests will be used for categorical variables, and independent t-tests for normally or Mann-Whitney U-test for non-normally distributed continuous variables. Generalized Linear Mixed Modelling (GLMM) will be employed for analyses of most outcome, except for the analyses of time to reabuse (part of research question 1) and time to premature termination (part of research question 5). For those outcomes, survival analysis (Cox regression) will be used.

ELIGIBILITY:
CRITERIA AT START (n = 11 included according to):

Inclusion Criteria:

* At least one adult residing in the family is suspected to have perpetrated an abusive act towards a child.
* The social services has decided to start a formal investigation of the suspected act.
* At least one child in the family is between 3 and 12 years old.

Exclusion Criteria:

* The social services already has an ongoing intervention with the family at the time when the suspected act is reported.

REVISED CRITERIA (n = 101 included according to):

Criteria were specified at beginning of inclusion (early spring 2020) to ensure that the intended population of Safer Kids could be recruited.

Revised inclusion criteria:

1. At least one adult in the family is suspected to have perpetrated an abusive act towards a child, resulting in an initiated child welfare investigation.
2. The suspected adult lives with the child, at least part time, during the investigation
3. At least one child in the family is between 2-12 years old.

Revised exclusion criteria:

1. The events preceding the report does not concern the child between 2-12 years old, only a younger or older sibling
2. The participating caregivers have participated in an intervention concerning abuse of children at the social services in the past 12 months
3. Caregiver and focus child lack residence permit the coming 30 months
4. The family's problem are assessed to be so severe that there is great risk of out-of-home placement of the child during the investigation.

Ages: 2 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 112 (Actual)
Dates: Start 2019-11-15 (Actual); Primary Completion 2024-06-01 (Actual); Study Completion 2024-06-01 (Actual)

PRIMARY OUTCOMES:
Change in Brief Child Abuse Potential Inventory (B-CAP) | Pre (0 month), Post (4 month), Follow-up (7 month), long-term follow-up (18 and 30 month)
  A short version of the well established CAP, which measures empirically established risk-factors for child abuse. The short version includes 24 items.
Change in Journal records: further reports on abuse or violence | 4-months, 7-months, 18-months and 30-months from baseline.
  On four occasions, personnel at the included social services units will extract information from the participating families journal records. The data that will be collected by the research team is: number of additional reports to the social services concerning the family, the date of each report, as well as the reason for each report.

SECONDARY OUTCOMES:
Change in Parent Anger Scale (PAS) | Pre (0 month), Post (4 month) and Follow-up (7 month)
  An instrument that measures caregivers anger directed at their child. The instrument includes two subscales; experienced anger and expressed anger. In this study, only the first subscale will be used, since the second includes questions regarding violent acts towards children.
Change in Perceived stress scale (PSS) | Pre (0 month), Post (4 month) and Follow-up (7 month)
  The scale will be used to measure parental stress. This is a frequently used scale consisting of 10 items in this version, which measures perceived stress.
Change in Patient Health Questionnaire (PHQ-9) | Pre (0 month), Post (4 month) and Follow-up (7 month)
  The scale will be used to measure parental level of depression (9 items), which is a well known risk factor for child abuse.
Change in The Strength and Difficulties Questionnaire (SDQ) | Pre (0 month), Post (4 month), Follow-up (7 month), long-term follow-up (18 and 30 month)
  To measure the well-being of the child, the caregivers in the study will complete the SDQ - 20 items.
Change in Kindl-R | Pre (0 month), Post (4 month) and Follow-up (7 month)
  The children who participate in the study will be interviewed by the practitioner. The interviews are structured and based on the Kindl-R, which is a scale that the practitioner will help the child to complete. The scale measures quality of life and in this study a few subscales will be included (total 8 items).
Change in The Alabama Parenting Questionnaire | Pre (0 month), Post (4 month) and Follow-up (7 month)
  Seven items will be used to measure the quality of the relationship between the caregivers and the child. The scale will be administrated to the parents.
Change in The Adult Child Relationship Scale (ACRS) | Pre (0 month), Post (4 month) and Follow-up (7 month)
  Also this scale is rated by the caregivers and will be used to measure the quality of the relationship between the caregivers and the child. The sub-scale measuring the level of warmth in the relationship will be used.
Client Satisfaction Questionnaire (CSQ-8) | Follow-up (7 month)
  Caregivers rated CSQ-8 to assess satisfaction with the help they received from the social services.
Practitioner Acceptability Questionnaire | Follow-up (7 month)
  A 7-item instrument pertaining to satisfaction of interventions was developed by the research group and administered to social workers. The questions concerned social workers view on intervention quality and helpfulness. Items were rated on a 4 point likert-scale. If the family did not receive any services, a fifth option 'no support/interventions' were checked.
Change in AUDIT-C | Pre (0 month), Post (4 month) and Follow-up (7 month)
  A 3-item questionnaire concerning alcohol consumption. Parents rate both regarding their own habits and the child's other guardian.
Change in GAD-7 | Pre (0 month), Post (4 month) and Follow-up (7 month)
  A well-established 7-item instrument rated by parents to assess worry and/or anxiety.

OTHER OUTCOMES:
Safer Kids Manual Adherence Rating Scale | After completion of Safer Kids
  After completion of Safer Kids, therapists rate how well they were able to carry out the main parts of each Safer Kids-theme according to the manual. Questions are rated on a 5 point likert-scale (range from 'not at all/not completed' to 'completely according to the manual'). The questionnaire also includes a question of potential obstacles in adhering to the manual.
Therapist Background Survey | After starting or completing treatment with first study family
  Therapists treating families in the study answer a survey containing questions about their background and education. Therapists educated in Safer Kids also answer two questions pertaining to support from the organisation in working with the intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Martin Forster, PhD, Principal Investigator — Karolinska Institutet
Locations (30):
- Sweden (30):
  - Alingsås kommun, Alingsås, Alingsås
  - Bjuvs kommun, Bjuv, Bjuv
  - Danderyds kommun, Djursholm, Djursholm
  - Fagersta kommun, Fagersta, Fagersta
  - Gislaveds kommun, Gislaved, Gislaved
  - Gävle kommun, Gävle, Gävle
  - Hudiksvalls kommun, Hudiksvall, Hudiksvall
  - Hörby kommun, Hörby, Hörby
  - Höörs kommun, Höör, Höör
  - Katrineholms kommun, Katrineholm, Katrineholm
  - Lerums kommun, Lerum, Lerum
  - Luleå kommun, Luleå, Luleå
  - Mönsterås kommun, Mönsterås, Mönsterås
  - Skara kommun, Skara, Skara
  - Skellefteå kommun, Skellefteå, Skellefteå
  - Staffanstorps kommun, Staffanstorp, Staffanstorp
  - Stenungsunds kommun, Stenungsund, Stenungsund
  - Sundbybergs stad, Sundbyberg, Sundbyberg
  - Sundsvalls kommun, Sundsvall, Sundsvall
  - Söderhamns kommun, Söderhamn, Söderhamn
  - Södertälje kommun, Södertälje, Södertälje
  - Tidaholms kommun, Tidaholm, Tidaholm
  - Botkyrka kommun, Tumba, Tumba
  - Täby kommun, Täby, Täby
  - Uppsala kommun, Uppsala, Uppsala County
  - Vellinge kommun, Vellinge, Vellinge
  - Lidingö kommun, Lidingö
  - Ronneby kommun, Ronneby
  - Österåkers kommun, Åkersberga, Åkersberga
  - Örebro kommun, Örebro, Örebro County

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Annerback EM, Wingren G, Svedin CG, Gustafsson PA. Prevalence and characteristics of child physical abuse in Sweden - findings from a population-based youth survey. Acta Paediatr. 2010 Aug;99(8):1229-36. doi: 10.1111/j.1651-2227.2010.01792.x. Epub 2010 Mar 8. PMID 20219025
- [Background] Stoltenborgh M, Bakermans-Kranenburg MJ, van Ijzendoorn MH, Alink LR. Cultural-geographical differences in the occurrence of child physical abuse? A meta-analysis of global prevalence. Int J Psychol. 2013;48(2):81-94. doi: 10.1080/00207594.2012.697165. PMID 23597008
- [Background] Norman RE, Byambaa M, De R, Butchart A, Scott J, Vos T. The long-term health consequences of child physical abuse, emotional abuse, and neglect: a systematic review and meta-analysis. PLoS Med. 2012;9(11):e1001349. doi: 10.1371/journal.pmed.1001349. Epub 2012 Nov 27. PMID 23209385
- [Background] Euser S, Alink LR, Stoltenborgh M, Bakermans-Kranenburg MJ, van IJzendoorn MH. A gloomy picture: a meta-analysis of randomized controlled trials reveals disappointing effectiveness of programs aiming at preventing child maltreatment. BMC Public Health. 2015 Oct 18;15:1068. doi: 10.1186/s12889-015-2387-9. PMID 26476980
- [Background] Vlahovicova K, Melendez-Torres GJ, Leijten P, Knerr W, Gardner F. Parenting Programs for the Prevention of Child Physical Abuse Recurrence: A Systematic Review and Meta-Analysis. Clin Child Fam Psychol Rev. 2017 Sep;20(3):351-365. doi: 10.1007/s10567-017-0232-7. PMID 28378136
- [Background] Kling A, Forster M, Sundell K, Melin L. A randomized controlled effectiveness trial of parent management training with varying degrees of therapist support. Behav Ther. 2010 Dec;41(4):530-42. doi: 10.1016/j.beth.2010.02.004. Epub 2010 Oct 1. PMID 21035616
- [Background] Stattin H, Enebrink P, Ozdemir M, Giannotta F. A national evaluation of parenting programs in Sweden: The short-term effects using an RCT effectiveness design. J Consult Clin Psychol. 2015 Dec;83(6):1069-1084. doi: 10.1037/a0039328. Epub 2015 May 25. PMID 26009784
- [Background] Chen M, Chan KL. Effects of Parenting Programs on Child Maltreatment Prevention: A Meta-Analysis. Trauma Violence Abuse. 2016 Jan;17(1):88-104. doi: 10.1177/1524838014566718. Epub 2015 Jan 8. PMID 25573846
- [Background] Lundahl BW, Nimer J, Parsons B. Preventing Child Abuse: A Meta-Analysis of Parent Training Programs. Research on Social Work Practice, 16(3): 251-262, doi: 10.1177/1049731505284391. Epub 2006.
- [Background] Faul F, Erdfelder E, Buchner A, Lang AG. Statistical power analyses using G*Power 3.1: tests for correlation and regression analyses. Behav Res Methods. 2009 Nov;41(4):1149-60. doi: 10.3758/BRM.41.4.1149. PMID 19897823
- [Derived] van Leuven L, Enebrink P, Ghaderi A, Sorjonen K, Lalouni M, Forster M. A randomized controlled trial of Safer Kids - A program for parents reported for child abuse: Short-term effects on further reports of child abuse and related risk factors. Child Abuse Negl. 2023 Sep;143:106329. doi: 10.1016/j.chiabu.2023.106329. Epub 2023 Jun 27. PMID 37384960